CLINICAL TRIAL: NCT07037823
Title: Effectiveness of the Combination Strategy of Disease-Modifying Therapy and the Yishen Daluo Yin Modified Formula for Multiple Sclerosis: A Prospective Multi-Center Observational Comparative Study
Brief Title: Effectiveness of the Combination Strategy of Disease-Modifying Therapy and the Yishen Daluo Yin Modified Formula for Multiple Sclerosis
Status: Not yet recruiting | Type: Observational
Sponsor: Ying Gao (Other)
Collaborators: The Second Hospital of Hebei Medical University (Other); First Affiliated Hospital of Jinan University (Other); Chinese PLA General Hospital (Other)
Responsible Party: Sponsor-Investigator, Ying Gao, Professior, Dongzhimen Hospital, Beijing
Organization: Dongzhimen Hospital, Beijing (Other)
Other Study IDs: 2024DZMEC-605
Record Dates: First submitted 2025-06-09; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-05

CONDITIONS: RRMS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DMT group: RRMS patients receiving DMT.
- YSDLY group: RRMS patients receiving DMT combining modified YSDLY formula.
  Interventions: Other: Modified Yishen Daluo Yin formula

INTERVENTIONS:
Other: Modified Yishen Daluo Yin formula — The specific application of the modified Yishen Daluo Yin formula, including the starting point, dosage, and duration of treatment, should be determined based on medical advice, the patient's condition, and their individual preferences.
  Groups: YSDLY group

SUMMARY:
This study was designed to investigate the effectiveness of a combined strategy utilizing disease-modifying therapy and the modified Yishen Daluo Yin formula for relapsing-remitting multiple sclerosis (RRMS) through a prospective, multicenter, observational comparative study.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who are over 18 years old at the time of signing the informed consent form, with no gender restrictions.
2. Participants meet the diagnostic criteria for multiple sclerosis (MS) as outlined in the 2017 McDonald's diagnostic criteria and the 2023 edition of the Chinese Guidelines for the Diagnosis and Treatment of Multiple Sclerosis.
3. No clinical relapse, as defined in the protocol, has occurred for 30 days or more prior to screening and baseline (Day 1).
4. Patients receiving first-line DMT drug treatment at a stable dosage. (The first-line DMT drugs involved in this study have stable dosages: Teriflunomide (14 mg, oral, once daily), Dimethyl Fumarate (240 mg, oral, twice daily), Fingolimod Hydrochloride (0.5 mg, oral, once daily), Siponimod (1 mg or 2 mg daily), Ozanimod (0.92 mg, oral, once daily), Ofatumumab (20 mg, subcutaneous injection once every 28 days), and Glatiramer Acetate (20 mg, subcutaneous injection once daily or 40 mg, three times a week).)
5. Signing the informed consent form.
6. Participants were able to engage in clinical follow-up throughout the entire study period.

Exclusion Criteria:

1. According to the 2017 McDonald's guidelines and the 2023 version of the Chinese Multiple Sclerosis Diagnosis and Treatment Guidelines, individuals diagnosed with progressive MS, including both primary progressive MS (PPMS) and secondary progressive MS (SPMS), are excluded.
2. Participants who cannot performe MRI scans in certain situations include individuals with known allergic reactions to gadolinium contrast agents or those with other contraindications.
3. The expected lifespan is less than one year.
4. Participants who cannot complet the study due to mental illness, cognitive or emotional disorders.
5. Pregnant or lactating women.
6. Patients who are currently receiving or participating in other immunosuppressive, immunomodulatory, MS DMT treatment or clinical trials.
7. Any situation that other researchers deem inappropriate for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a multicenter study, participants are from Beijing, Hebei, and Guangzhou.
Sampling Method: Probability Sample
Enrollment: 328 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients exhibiting no evidence of disease activity (NEDA) -3 at 48 weeks. | From enrollment to week 48.

SECONDARY OUTCOMES:
Annual Relapse Rate | From enrollment to week 24 and week 48.
Proportion of Patients Without Relapse | From enrollment to week 12, 24, 36, and 48.
Changes in EDSS Compared to Baseline | From enrollment to week 12, 24, 36, and 48.
The proportion of patients with confirmed disability progression within 3 months. | From enrollment to week 12, 24, 36, and 48.
The proportion of patients with confirmed disability progression within 6 months. | From enrollment to week 24 and week 48.
Number of newly added gadolinium enhanced T1 lesions | From enrollment to week 48.
Total number of gadolinium-enhanced T1 lesions | From enrollment to week 48.
Changes in T1 lesion volume compared with baseline | From enrollment to week 24 and week 48.
Number of newly added or enlargement gadolinium enhanced T2 lesions. | From enrollment to week 24 and week 48.
Changes in T2 lesion volume compared with baseline | From enrollment to week 24 and week 48.
Proportion of patients with treatment interruption | From enrollment to week 12, 24, 36, and 48.
Proportion of patients who terminated treatment | From enrollment to week 12, 24, 36, and 48.
Proportion of patients who switch treatments | From enrollment to week 12, 24, 36, and 48.

IPD SHARING:
Plan to Share IPD: No